CLINICAL TRIAL: NCT03709446
Title: A Phase I/II Trial of Leflunomide in Women With Previously Treated Metastatic Triple Negative Cancers
Brief Title: Leflunomide in Previously Treated Metastatic Triple Negative Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph Sparano (Other)
Responsible Party: Sponsor-Investigator, Joseph Sparano, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1832
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; Breast Diseases; Metastatic Triple Negative Breast Cancer
Keywords: Breast Neoplasms; Breast Diseases; Leflunomide; Teriflunomide; Phosphatase and tensin homolog
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Triple Negative Breast Neoplasms | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leflunomide (Experimental): Women with HER2-negative metastatic and/or locally advanced, inoperable breast cancer.
  Leflunomide tablet orally daily
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Single agent leflunomide
  Other Names: Arava

SUMMARY:
Triple negative breast cancer (TNBC) represents about 15% of breast cancers and is characterized by the lack of expression of estrogen receptor (ER), progesterone receptor (PR), and HER-2 non-amplification. Women with TNBC tend to be younger, African American, and BRCA-1 germline carriers. The hallmark of this subtype is early metastatic recurrences with a peak frequency 1-2 years. Prognosis for metastatic TNBC is especially poor with median survival of about 1 year as compared to about 2-4 years with other types of metastatic breast cancer.

The primary objective of the phase I part of this study is to determine the safety, tolerability and maximum tolerated dose of leflunomide in women with previously treated TNBC (or ER+ , HER2-neg MBC in Phase I). The primary objective of the phase 2 part of this study is to determine the efficacy of leflunomide in patients with TNBC.

Leflunomide, which will be taken daily by mouth, is an inhibitor of dihydroorotate dehydrogenase (DHODH). This proposal will test if DHODH is a novel target for a particular subset of women with metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed HER2-negative metastatic and/or locally advanced, inoperable breast cancer on a prior biopsy performed as a component of standard of care. The biopsy site may include the primary tumor, regional lymph node, or metastatic site if accessible to biopsy.
* Age ≥ 18.
* Prior treatment for metastatic breast cancer:
* ≤ 3 prior chemotherapies for metastatic disease and up to 2 prior antibody drug conjugate regimens (eg, sacitizumab govitecan, trastuzumab deruxtecan). Patients with ER-positive breast cancer (ER>10%) must have had progressive disease after at least 1 prior line of CKD4/6 inhibitor, and also a PIK3CA inhibitor if known to have a somatic PIK3CA activating mutation (by tumor or ctDNA assay) sensitive to the PIK3CA inhibitor alpelisib.
* Prior immunotherapy is permitted and does not count as chemotherapy.
* The use denosumab or zoledronic is permitted.
* History of previously treated brain metastases with ≥ 4 weeks after definitive surgery and gamma knife/whole brain radiation and not taking steroids.
* ≥ 4 weeks from last oral or IV chemotherapy, small molecule inhibitor, a biologic agent, surgery or radiation.
* Performance status 0-2.
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 100,000/mcl
  * total bilirubin within institutional upper limit of normal. (≤ ULN)
  * AST (SGOT)/ALT (SPGT) ≤ 3 x ULN (3xULN if liver mets)
  * Creatinine ≤ ULN
  * A negative serum or urine pregnancy test within 3 days of receiving Day 1 Cycle 1 of leflunomide.
* Women of child-bearing potential and men must agree to use adequate contraception before study entry, for the duration of study participation and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Recommended methods of birth control are: The consistent use of an approved hormonal contraception such as an intrauterine device (IUD), Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam), Sexual abstinence (no sexual intercourse) or Sterilization. The use of hormonal forms of birth control is controversial in TNBC and as such women enrolled in the trial are permitted to use birth control pills or depot Provera, only after a documented discussion by the treating physician as too the uncertain risks of hormonal birth control methods in the TNBC population. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within ≥ 2 weeks before entering the study or those who have not recovered from adverse events due to agents administered more than ≥ 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* The known history human immunodeficiency virus, acute and chronic Hepatitis B or C, or acute or previously treated tuberculosis.
* Patients with untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leflunomide or teriflunomide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 months
  3+3 escalation schema. Patients will be enrolled in escalating cohorts of 3 patients per dose level until Dose-limiting Toxicity (DLT) (defined as any grade 3 or higher toxicity seen during the first 3-week cycle of leflunomide). If 0 of 3 patients are observed to have a DLT, the next 3 patients will be enrolled in the next higher dose level cohort. If 2/3 patients experience a DLT, escalation will stop and the previous dose will be defined as the MTD. If 1/3 experiences a DLT, three additional patients will be enrolled at the same dose level. If ≤ 2/6 patients experience a DLT, the next cohort of three patients will be treated at the next dose level. If ≥ 3/6 experience a DLT, the next lower dose level will define the MTD. If at the 50 mg dose/day if 0/3 or ≤ 2/6 patients experience a DLT, then that dose will define the MTD
Clinical Benefit Rate (CBR) | 6 months
  Response and progression to be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST). CBR = Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) for at least 6 months duration

SECONDARY OUTCOMES:
Number of side effects | 6 years
  Number of side effects associated with oral leflunomide using NCI CTCAE v.4.03
Objective Response Rate | 6 years
  Objective Response Rate (proportion of patients with the best overall response of CR or PR) in those who have measurable disease by RECIST
Progression-free survival (PFS) | 6 years
  PFS of women with phosphatase and tensin homolog (PTEN) wild-type and PTEN null expression breast cancers. PFS is defined as the duration of time from the start of treatment to the first occurrence of disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mt Sinai Chelesa, New York, New York
  - Mt Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No